CLINICAL TRIAL: NCT02979184
Title: Prevalence of Obstructive Sleep Apnea Syndrom in Patients With Lymphedema, Admitted for Intensive Decongestive Physiotherapy
Brief Title: Prevalence of Obstructive Sleep Apnea (OSA) in Patients With Lymphedema, Admitted for Intensive Decongestive Physiotherapy
Acronym: LYMPHOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC16.204
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Lymphedema; Obstructive Sleep Apnea Syndrome
Keywords: Lymphedema, Obstructive Sleep Apnea , Intensive Decongestive Physiotherapy
MeSH Terms: conditions — Lymphedema; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensive decongestive physiotherapy (Other): 2 weeks of intensive decongestive physiotherapy
  Interventions: Other: Intensive decongestive physiotherapy

INTERVENTIONS:
Other: Intensive decongestive physiotherapy — 2 weeks of intensive decongestive physiotherapy

SUMMARY:
Rehabilitation results in a decrease of the perimeters of the limb with lymphedema by a decrease in the amount of liquid of the affected limb, with movement of the intracellular liquid towards the trunk and the neck then into the jugular-subclavian confluence, the superior vena cava and right atrium without modification of extracellular fluid. No study have evaluated the prevalence of sleep apnea syndrome in this population and the effect of this treatment on sleep apnea syndrome.

DETAILED DESCRIPTION:
Lymphedema is the result of an intra-tissue fluid accumulation by failure of the lymphatic system to absorb the excess fluid from the veinulo-capillary circulation. Lymphedema can be primitive with aplasia or hypoplasia of the lymphatic vessels or secondary by destruction of the lymphatic structures.

We define three stages of severity of lymphedema:

* Stage I: increase of volume which is mitigate when the limb is raised
* Stage II: the elevation does not reduce anymore the volume and the oedema is still compressible. It produces skin changes such as fibrosis, rendered by the sign of Stemmer.
* Stage III: elephantiasis with disappearance of the compressible nature of edema, appearance of trophic skin disorders (papillomas, vesicles) and nail disorders.

The first-line treatment of lymphedema corresponds to a physical therapy by decongestive physiotherapy. This intensive rehabilitation includes sessions of manual lymphatic drainages or pressure therapy sessions followed by the application of inelastic multilayer bandages, muscle exercises under bandages, skin care and pedicure for lymphedema of the lower limbs.

Rehabilitation results in a decrease of the perimeters of the limb with lymphedema by a decrease in the amount of liquid of the affected limb, with movement of the intracellular liquid towards the trunk and the neck then into the jugular-subclavian confluence, the superior vena cava and right atrium without modification of extracellular fluid. No study have evaluated the prevalence of sleep apnea syndrome in this population and the effect of this treatment on sleep apnea syndrome.

The interest of this study is to evaluate the prevalence of sleep apnea syndrome at patients suffering from lymphedema and the effect of intensive decongestive physiotherapy on the syndrome of sleep apnea by modification of the fluid redistribution.

ELIGIBILITY:
Inclusion Criteria:

* Lymphedema of one or several limbs (with difference of more than 2 cms compared with the collateral limb) without contraindication in an intensive decongestive physiotherapy.
* Patient member to the social security or beneficiary of such a regime.
* Patient having signed the informed consent for participation to the study

Exclusion Criteria:

* Medical Contraindication in an intensive decongestive physiotherapy : Acute infectious episode (Erysipelas, lymphangitis), acute venous thrombosis, uncontrolled heart failure or hypertension, acute renal failure, obstruction of the superior vena cava, evolutionary untreated malignant tumor, peripheral arterial disease with ankle brachial indices w< 0,5, evolved diabetic angiopathy, septic thrombosis, popliteal aneurysm.
* Patients deprived of freedom by court or admninistrative order. Person being the object of a legal protective measure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea syndrom in patients with lymphedema, admitted for intensive decongestive physiotherapy. | 1 year
  Apnea/hypopnea index (AHI /h) measured by Apnea-Link or antecedent of Obstructive sleep apnea syndrom already treated with CPAP (Continuous Positive Airway Pressure) ventilation

SECONDARY OUTCOMES:
Effect of intensive decongestive physiotherapy on the severity of the obstructive sleep apnea syndrom of patients with apnea/hypopnea index ≥ 5 | 1 year
  Apnea/hypopnea index (AHI / h) before and after intensive decongestive physiotherapy.
Evolution of clinical signs associated with sleep apnea after rehabilitation | 1 year
  Clinical signs associated with sleep apnea: snoring, feeling of suffocation or oppression during sleep, non-restorative sleep, daytime fatigue, concentration difficulties, nocturia (clinical questionnaire)
Correlation between the volume of lymphedema of the suffering limb and the apnea/hypopnea index. | 1 year
  Measurement of limb perimeters (volumetry) before and after rehabilitation
Correlation between sleepiness measured by the Epworth scale before and after therapy, and the change in volume of lymphedema. | 1 year
  Score of the Epworth sleepiness scale before and after rehabilitation
Correlation between the quality of life as measured by the Medical Outcome Study Short Form questionnaire before and after rehabilitation, and apnea/hypopnea index. | 1 year
  Score in the MOS-SF-36 questionnaire before and after rehabilitation
Correlation between BMI (Body Mass Index) and apnea/hypopnea index. | 1 year
  BMI (kg/m^2)before and after rehabilitation
Correlation between perimeter of the neck and apnea/hypopnea index | 1 year
  Neck circumference (cm) before and after rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice VILLEMUR, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHUGA, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roux C, Villemur B, Giovannoni B, Koeyemelk L, Mendelson M, Benmerad M, Joyeux-Faure M, Tamisier R, Pepin JL. Prevalence of obstructive sleep apnea syndrome in patients with lymphedema referred for complete decongestive therapy. J Vasc Surg Venous Lymphat Disord. 2020 Jan;8(1):137-142. doi: 10.1016/j.jvsv.2019.07.007. Epub 2019 Oct 18. PMID 31636050